CLINICAL TRIAL: NCT02799069
Title: A Randomized, Observer Blind, Multinational Phase III Study to Evaluate the Safety and Efficacy of a Nanoemulsion Gel Formulation BF-200 ALA, in Comparison With Metvix® and Placebo, for the Treatment of Actinic Keratosis With PDT
Brief Title: Evaluation of Safety and Efficacy of BF-200 ALA for the Treatment of Actinic Keratosis With Photodynamic Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biofrontera Bioscience GmbH (Industry)
Collaborators: Accovion GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALA-AK-CT002
Record Dates: First submitted 2016-05-26; First posted 2016-06-14 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — BF-200 ALA; Aminolevulinic Acid; methyl 5-aminolevulinate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BF-200 ALA (Active Comparator): Topical application of BF-200 ALA gel containing 78 mg/g 5-aminolevulinic acid (ALA). Application of a 1 mm thick layer covering each lesion and a 0.5 cm to 1 cm surrounding margin.
  Interventions: Drug: BF-200 ALA
- MAL Cream (Active Comparator): Topical application of MAL cream (Metvix) containing 160 mg/g methyl-aminolevulinate (MAL). Application of a 1 mm thick layer covering each lesion and a 0.5 cm to 1 cm surrounding margin.
  Interventions: Drug: MAL Cream
- Vehicle (Placebo Comparator): Topical application of matched Placebo to BF-200 ALA gel (without containing active ingredient) ). Application of a 1 mm thick layer covering each lesion and a 0.5 cm to 1 cm surrounding margin.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: BF-200 ALA — topical treatment for photodynamic therapy combining drug application and after a 3 h incubation subsequent illumination with a broad or narrow spectrum light source.
  Other Names: Ameluz
  Arms: BF-200 ALA
Drug: MAL Cream — topical treatment for photodynamic therapy combining drug application and after a 3 h incubation subsequent illumination with a broad or narrow spectrum light source.
  Other Names: Metvix; Metvixia
  Arms: MAL Cream
Drug: Vehicle — topical treatment for photodynamic therapy combining vehicle application and after a 3 h incubation subsequent illumination with a broad or narrow spectrum light source.
  Other Names: matched placebo to BF-200 ALA gel
  Arms: Vehicle

SUMMARY:
The aim of the study is to evaluate the non-inferiority of BF-200 ALA (Ameluz) in the treatment of actinic keratosis (AK) with photodynamic therapy (PDT) compared to Metvix.

DETAILED DESCRIPTION:
This was a randomized, observer-blind, multinational, comparator and placebo-controlled parallel group, (3:3:1 ratio) study to compare the efficacy and safety of BF-200 ALA with the comparator Metvix® (methyl-[5-amino-4-oxopentanoate]) and placebo, for the treatment of AK with PDT.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent.
* Men and women between 18 and 85 years of age.
* 4-8 AK lesions of 0.5 to 1.5 cm diameter of mild to moderate intensity (Olsen grade 1 and 2) in the face and/or on the bald scalp. Lesions on the eyes, nostrils, ears and mouth were not considered for treatment during the planned study.
* Target AK lesions were to be discrete and quantifiable; adjacent AK lesions were to show a minimum distance of 1.0 cm from one another.
* Confirmation of AK by biopsy taken at screening.
* Free of significant physical abnormalities (e.g., tattoos, dermatoses) in the potential treatment region that could have caused difficulty with examination or final evaluation.
* Willingness to stop the use of moisturizers and any other topical treatments within the treatment region.
* Good general health condition.
* Healthy subjects and subjects with clinically stable medical conditions including, but not limited to the following diseases (controlled hypertension, diabetes mellitus type II, hypercholesterolemia, osteoarthritis) were permitted to be included in the study if the medication taken for the treatment of the disease did not match an exclusion criterion or was not specified as prohibited concomitant medication.
* No extensive sunbathing or solarium use during the trial.
* Negative pregnancy test at screening.

Main exclusion criteria:

* Known hypersensitivity to BF-200 ALA, MAL (methyl-aminolevulinic acid) and/or any of the ingredients of the formulations
* Clinically significant medical conditions (tumor disease etc.) making implementation of the protocol or interpretation of the study results difficult
* Presence of photodermatoses
* Presence of other tumors in the treatment areas within the last 4 weeks
* Start of treatment with phototoxic or photoallergic drugs within 8 weeks prior to screening
* Current treatment with immunosuppression therapy
* Hypersensitivity to porphyrins
* Presence of porphyria
* Presence of inherited or acquired coagulation defect
* Any topical treatment within the treatment area within 12 weeks before PDT1 (first PDT Treatment)
* Topical treatment with ALA or MAL outside the treatment area during participation in the study
* None of the specified systemic treatments within the designated period before PDT1

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dirschka, Prof. Dr., Principal Investigator — Akademische Lehrpraxis der Universität Witten-Herdecke Heinz-Fangman-Straße 57 42287 Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dirschka T, Radny P, Dominicus R, Mensing H, Bruning H, Jenne L, Karl L, Sebastian M, Oster-Schmidt C, Klovekorn W, Reinhold U, Tanner M, Grone D, Deichmann M, Simon M, Hubinger F, Hofbauer G, Krahn-Senftleben G, Borrosch F, Reich K, Berking C, Wolf P, Lehmann P, Moers-Carpi M, Honigsmann H, Wernicke-Panten K, Helwig C, Foguet M, Schmitz B, Lubbert H, Szeimies RM; AK-CT002 Study Group. Photodynamic therapy with BF-200 ALA for the treatment of actinic keratosis: results of a multicentre, randomized, observer-blind phase III study in comparison with a registered methyl-5-aminolaevulinate cream and placebo. Br J Dermatol. 2012 Jan;166(1):137-46. doi: 10.1111/j.1365-2133.2011.10613.x. Epub 2011 Dec 21. PMID 21910711
- [Background] Dirschka T, Radny P, Dominicus R, Mensing H, Bruning H, Jenne L, Karl L, Sebastian M, Oster-Schmidt C, Klovekorn W, Reinhold U, Tanner M, Grone D, Deichmann M, Simon M, Hubinger F, Hofbauer G, Krahn-Senftleben G, Borrosch F, Reich K, Berking C, Wolf P, Lehmann P, Moers-Carpi M, Honigsmann H, Wernicke-Panten K, Hahn S, Pabst G, Voss D, Foguet M, Schmitz B, Lubbert H, Szeimies RM; AK-CT002 Study Group; AK-CT003 Study Group. Long-term (6 and 12 months) follow-up of two prospective, randomized, controlled phase III trials of photodynamic therapy with BF-200 ALA and methyl aminolaevulinate for the treatment of actinic keratosis. Br J Dermatol. 2013 Apr;168(4):825-36. doi: 10.1111/bjd.12158. PMID 23252768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multinational / 26 centers sites: Germany (23), Austria (2) and Switzerland (1); 08 Apr 2008: First subject signed informed consent; 21 Aug 2009: Last subject completed clinical part of study
Pre-assignment Details: 616 patients with actinic keratosis (AK) were planned to be randomized in a 3:3:1 ratio allowing for 20% of non-evaluable patients excluded from the per-protocol set. Due to the low drop out rates, recruiting was stopped after 600 patients were screened. Of those, 571 patients were randomized and 29 patients were screening failures.
Groups:
- Vehicle: Topical application of BF-200 ALA matched placebo gel without active ingredient. Application of a 1 mm thick layer covering each lesion and a 0.5 cm to 1 cm surrounding margin.
  BF-200 ALA matched placebo: topical treatment for photodynamic therapy combining vehicle application and after a 3 h incubation subsequent illumination with a broad or narrow spectrum light source.
- MAL Cream: Topical application of MAL cream (Metvix) containing 160 mg/g methyl-aminolevulinate (MAL). Application of a 1 mm thick layer covering each lesion and a 0.5 cm to 1 cm surrounding margin.
  MAL: topical treatment for photodynamic therapy combining drug application and after a 3 h incubation subsequent illumination with a broad or narrow spectrum light source.
Period: Overall Study
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Started (randomized) | 76 | 248 | 247
ITT/Safety | 76 | 248 | 246 (1 subject received medication without Illumination and thus was excluded from ITT/safety population)
Completed | 68 | 241 | 240
Not Completed | 8 | 7 | 7
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 3
Not completed — Protocol Violation | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intended-to-treat (ITT)
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | BF-200 ALA | MAL Cream | Total
Number analyzed (Participants) | 76 | 248 | 246 | 570
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 47 | 38 | 94
  >=65 years | 67 | 201 | 208 | 476
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (6.68) | 70.2 (7.18) | 71.0 (6.93) | 70.7 (7.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 34 | 41 | 91
  Male | 60 | 214 | 205 | 479
Region of Enrollment [Number; unit: participants]
  Europe | 76 | 248 | 246 | 570
Number of individual lesions [Number; unit: individual lesions] | 490 | 1504 | 1557 | 3551

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response 12 Weeks After the Last Photodynamic Therapy (PDT), ITT
Description: An overall complete responder was defined as a subject in whom all treated lesions were cleared (all lesions showing complete remission) 12 weeks after the last PDT.
  The outcome measure considered complete responders who were completely cleared 12 weeks after the first PDT and responders who were completely cleared 12 weeks after the second PDT if a re-treatment was necessary (in case of partial- or non-responding lesions 12 weeks after the first PDT)
Time Frame: 12 weeks after the last PDT, up to 24 weeks after the first treatment
Population: Intent-to-treat (ITT)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
percentage of patients | 17.1 [9.4 to 27.5] | 78.2 [72.6 to 83.2] | 64.2 [57.9 to 70.2]
Statistical Analysis 1: Comparison: BF-200 ALA vs MAL Cream; Test type: Non-Inferiority — The sample size of 210 subjects per treatment arm (per protocol set) has a power of at least 90% to establish non-inferiority of BF-200 ALA to Metvix using a non-inferiority margin of -15% and assuming response rates of 70% for both BF-200 ALA and Metvix. The power calculation was based on a one-sided Z-test with continuity correction (unpooled) with a significance level of 0.025.The establishment of non-inferiority was performed for the PP set and verified for robustness on the ITT; Difference to BF-200 ALA = 14.0, 97.5% CI 1-sided [lower limit 5.9]
Statistical Analysis 2: Comparison: Vehicle vs BF-200 ALA; Superiority of BF-200 ALA compared to placebo: A sample size of 264: 88 patients (BF-200 ALA: placebo) will have a power of more than 90% to establish superiority of BF-200 ALA over placebo, even if very conservative response rates of 65% for the BF-200 ALA group and 40% for placebo are assumed using a chi-square test with continuity correction and a two-sided significance level of 0.05; Test type: Superiority; p = 0.0000, Chi-squared; Difference to BF-200 ALA = 61.1, 95% CI 2-sided [51.2 to 71.0]

2. Primary Outcome: Percentage of Participants With Complete Response 12 Weeks After the Last Photodynamic Therapy (PDT), PP
Description: as for outcome 1
Time Frame: 12 weeks after the last PDT, up to 24 weeks after the first treatment
Population: per protocol set (PP)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 65 | 238 | 236
percentage of patients | 20.0 [11.1 to 31.8] | 79.4 [73.7 to 84.4] | 65.3 [58.8 to 71.3]
Statistical Analysis 1: Comparison: BF-200 ALA vs MAL Cream; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference to BF-200 ALA = 14.2, 97.5% CI 1-sided [lower limit 6.0]
Statistical Analysis 2: Comparison: Vehicle vs BF-200 ALA; Test type: Superiority or Other; p = 0.0000, Chi-squared; Difference to BF-200 ALA = 59.4, 95% CI 2-sided [48.4 to 70.4]

3. Primary Outcome: Percentage of Participants With Complete Response 12 Weeks After the Last Photodynamic Therapy (PDT) Illuminated With Narrow Spectrum Devices Only
Description: Subgroup analysis of patients treated with a narrow spectrum device for PDT Illumination (~630 nm).
  An overall complete responder was defined as a subject in whom all treated lesions were cleared (all lesions showing complete remission) 12 weeks after the last PDT.
  The outcome measure considered complete responders who were completely cleared 12 weeks after the first PDT and responders who were completely cleared 12 weeks after the second PDT if a re-treatment was necessary (in case of partial- or non-responding lesions 12 weeks after the first PDT)
Time Frame: 12 weeks after the last PDT, up to 24 weeks after the first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 39 | 125 | 126
percentage of patients | 12.8 [4.3 to 27.4] | 84.8 [77.3 to 90.6] | 67.5 [58.5 to 75.5]
Statistical Analysis 1: Comparison: Vehicle vs BF-200 ALA; Test type: Superiority or Other; p = 0.0000, Chi-squared; Difference to BF-200 ALA = 72.0, 95% CI 2-sided [59.7 to 84.2]
Statistical Analysis 2: Comparison: BF-200 ALA vs MAL Cream; Test type: Superiority or Other; Difference to BF-200 ALA = 17.3, 97.5% CI 1-sided [lower limit 6.6]

4. Secondary Outcome: Percentage of Participants With Complete Response 3-4 Weeks After First Photodynamic Therapy (PDT)
Description: A complete responder was defined as a subject in whom all treated lesions were cleared (all lesions showing complete remission) at 3-4 weeks after the first PDT.
Time Frame: 3-4 weeks after the first PDT
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
percentage of patients | 2.6 [0.3 to 9.2] | 34.7 [28.8 to 41.0] | 24.8 [19.5 to 30.7]

5. Secondary Outcome: Percentage of Participants With Complete Response 12 Weeks After First Photodynamic Therapy (PDT)
Description: A complete responder was defined as a subject in whom all treated lesions were cleared (all lesions showing complete remission) at 12 weeks after the first PDT.
Time Frame: 12 weeks after the first PDT
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
percentage of patients | 3.9 [0.8 to 11.1] | 48.4 [42.0 to 54.8] | 37.0 [30.9 to 43.4]

6. Secondary Outcome: Percentage of Participants With Complete Response 3-4 Weeks After the Second Photodynamic Therapy (PDT)
Description: A complete responder was defined as a subject in whom all treated lesions were cleared (all lesions showing complete remission) at 3-4 weeks after the second PDT. A second PDT was applied in case partial- or non-responding lesions remained 12 weeks after the first PDT.
Time Frame: 3-4 weeks after the second PDT, 15-16 weeks after first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 73 | 128 | 155
percentage of patients | 13.7 [6.8 to 23.8] | 48.4 [39.5 to 57.4] | 43.9 [35.9 to 52.1]

7. Secondary Outcome: Percentage of Participants With Complete Response 12 Weeks After Second Photodynamic Therapy (PDT)
Description: A complete responder was defined as a subject in whom all treated lesions were cleared (all lesions showing complete remission) at 12 weeks after the second PDT. A second PDT was applied in case partial- or non-responding lesions remained 12 weeks after the first PDT.
Time Frame: 12 weeks after the second PDT, 24 weeks after first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 73 | 128 | 155
percentage of patients | 13.7 [6.8 to 23.8] | 57.8 [48.8 to 66.5] | 43.2 [35.3 to 51.4]

8. Secondary Outcome: Percentage of Participants With Complete Response 3-4 Weeks After Last Photodynamic Therapy (PDT)
Description: A complete responder at week 3-4 after treatment was defined as a subject in whom all treated lesions were cleared (all lesions showing complete remission). This outcome measure considered patients who were completely cleared at 3-4 weeks after the last PDT which included complete responders 3-4 weeks after the first and complete responders 3-4 weeks after the second PDT ( a second PDT was applied in case of remaining lesions 12 weeks after the first PDT).
Time Frame: 3-4 weeks after the last PDT, up to 16 weeks after the first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
percentage of patients | 14.5 [7.5 to 24.4] | 54.0 [47.6 to 60.4] | 43.9 [37.6 to 50.3]

9. Secondary Outcome: Percentage of Participants With Partial Response at 3-4 Weeks After First Photodynamic Therapy (PDT)
Description: A partial responder was defined as a subject in whom at least 75% of the treated lesions were cleared (lesions showing complete remission). This outcome measure considers partial responders at 3-4 weeks after the first PDT.
Time Frame: 3-4 weeks after the first PDT
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
percentage of patients | 2.6 [0.3 to 9.2] | 50.0 [43.6 to 56.4] | 45.9 [39.6 to 52.4]

10. Secondary Outcome: Percentage of Participants With Partial Response at 12 Weeks After the First Photodynamic Therapy (PDT)
Description: A partial responder was defined as a subject in whom at least 75% of the treated lesions were cleared (lesions showing complete remission). This outcome measure considers partial responders at 12 weeks after the first PDT.
Time Frame: 12 weeks after the first PDT
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
percentage of patients | 13.2 [6.5 to 22.9] | 58.9 [52.5 to 65.1] | 53.3 [46.8 to 59.6]

11. Secondary Outcome: Percentage of Participants With Partial Response at 3-4 Weeks After the Second Photodynamic Therapy (PDT)
Description: A partial responder was defined as a subject in whom at least 75% of the treated lesions were cleared (lesions showing complete remission). This outcome measure considers partial responders at 3-4 weeks after the second PDT.
  A second PDT was applied in case of partial- or non-responding lesions 12 weeks after the first PDT.
Time Frame: 3-4 weeks after the second PDT, 15-16 weeks after first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 73 | 128 | 155
percentage of patients | 20.5 [12.0 to 31.6] | 68.0 [59.1 to 75.9] | 62.6 [54.5 to 70.2]

12. Secondary Outcome: Percentage of Participants With Partial Response at 12 Weeks After the Second Photodynamic Therapy (PDT)
Description: A partial responder was defined as a subject in whom at least 75% of the treated lesions were cleared (lesions showing complete remission). This outcome measure considers partial responders at 12 weeks after the second PDT.
  A second PDT was applied in case of partial- or non-responding lesions 12 weeks after the first PDT.
Time Frame: 12 weeks after the second PDT, 24 weeks after first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 73 | 128 | 155
percentage of patients | 23.3 [14.2 to 34.6] | 73.4 [64.9 to 80.9] | 65.2 [57.1 to 72.6]

13. Secondary Outcome: Percentage of Participants With Partial Response at 3-4 Weeks After Last Photodynamic Therapy (PDT)
Description: A partial responder was defined as a subject in whom at least 75% of the treated lesions were cleared (lesions showing complete remission). This outcome measure considers partial responders at 3-4 weeks after last PDT.
  The outcome measure combined partial responders with at least 75% of lesions cleared at 3-4 weeks after the first PDT or after the second PDT (a second PDT was applied in case of partial- or non-responding lesions 12 weeks after the first PDT).
Time Frame: 3-4 weeks after the last PDT, up to 16 weeks after the first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
percentage of patients | 21.1 [12.5 to 31.9] | 70.6 [64.5 to 76.2] | 64.6 [58.3 to 70.6]

14. Secondary Outcome: Percentage of Participants With Partial Response at 12 Weeks After Last Photodynamic Therapy (PDT)
Description: A partial responder was defined as a subject in whom at least 75% of the treated lesions were cleared (lesions showing complete remission). This outcome measure considers partial responders at 12 weeks after last PDT.
  The outcome measure combined partial responders with at least 75% of lesions cleared at 12 weeks after the first PDT and after the second PDT (a second PDT was applied in case of partial- or non-responding lesions 12 weeks after the first PDT) .
Time Frame: 12 weeks after the last PDT, up to 24 weeks after first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
percentage of patients | 26.3 [16.9 to 37.7] | 87.1 [82.3 to 91.0] | 78.0 [72.3 to 83.1]

15. Secondary Outcome: Complete Lesion Response Rate 3-4 Weeks After First Photodynamic Therapy (PDT)
Description: Completely cleared individual lesions as defined at 3-4 weeks after first photodynamic therapy (PDT)
Time Frame: 3-4 weeks after the first PDT
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: number of individual lesions
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
Number analyzed (number of individual lesions) | 490 | 1504 | 1557
percentage of lesions | 12.7 [9.8 to 15.9] | 63.9 [61.4 to 66.3] | 58.8 [56.3 to 61.3]

16. Secondary Outcome: Complete Lesion Response Rate 12 Weeks After First Photodynamic Therapy (PDT)
Description: Completely cleared individual lesions as defined at 12 weeks after the first photodynamic therapy (PDT).
Time Frame: 12 weeks after the first PDT
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: number of individual lesions
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
Number analyzed (number of individual lesions) | 490 | 1504 | 1557
percentage of lesions | 24.7 [20.9 to 28.8] | 73.8 [71.5 to 76.0] | 66.5 [64.1 to 68.8]

17. Secondary Outcome: Complete Lesion Response Rate 3-4 Weeks After the Second Photodynamic Therapy (PDT)
Description: Completely cleared individual lesions as defined at 3-4 weeks after the second PDT. A second PDT was applied in case the individual lesion showed no or partial response12 weeks after first PDT.
Time Frame: 3-4 weeks after the second PDT, 15-16 weeks after first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: number of individiual lesions
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 73 | 128 | 155
Number analyzed (number of individiual lesions) | 369 | 394 | 522
percentage of lesions | 16.3 [12.6 to 20.4] | 60.4 [55.4 to 65.3] | 54.8 [50.4 to 59.1]

18. Secondary Outcome: Complete Lesion Response Rate 12 Weeks After Second PDT
Description: Completely cleared individual lesions as defined at 12 weeks after second PDT. A second PDT was applied in case the individual lesion showed no or partial response 12 weeks after first PDT.
Time Frame: 12 weeks after the second PDT, 24 weeks after first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: number of individual lesions
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 73 | 128 | 155
Number analyzed (number of individual lesions) | 369 | 394 | 522
percentage of lesions | 22.0 [17.8 to 26.5] | 69.3 [64.5 to 73.8] | 58.0 [53.7 to 62.3]

19. Secondary Outcome: Complete Lesion Response Rate 3-4 Weeks After Last Photodynamic Therapy (PDT)
Description: Completely cleared individual lesions defined at 3-4 weeks after the last PDT comprising of completely cleared individual lesions 3-4 weeks after the first and after the second PDT (a second PDT was applied in case lesions show no or partial response 12 weeks after the first PDT).
Time Frame: 3-4 weeks after the last PDT, up to 16 weeks after first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: number of individual lesions
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
Number analyzed (number of individual lesions) | 490 | 1504 | 1557
percentage of lesions | 31.4 [27.3 to 35.7] | 79.0 [76.8 to 81.0] | 73.5 [71.2 to 75.7]

20. Secondary Outcome: Complete Lesion Response Rate 12 Weeks After Last Photodynamic Therapy (PDT)
Description: Completely cleared individual lesions 12 weeks after last PDT comprising of completely cleared individual lesions 12 weeks after the first or second PDT (a second PDT was applied in case individual lesions show no or partial response 12 weeks after first PDT).
Time Frame: 12 weeks after the last PDT, up to 24 weeks after first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: num,ber of individual lesions
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
Number analyzed (num,ber of individual lesions) | 490 | 1504 | 1557
percentage of lesions | 37.1 [32.9 to 41.6] | 90.4 [88.8 to 91.8] | 83.2 [81.2 to 85.0]

21. Secondary Outcome: Complete Lesion Response Rates 12 Weeks After Last Photodynamic Therapy (PDT) Illuminated With Narrow Spectrum Devices Only
Description: Completely cleared individual lesions 12 weeks after last PDT comprising of individual cleared lesions 12 weeks after the first or second PDT. A second PDT was applied in case individual lesion showed no or partial response 12 weeks after the first PDT.
  Lesions were illuminated during photodynamic therapy with narrow spectrum devices only (~630 nm).
Time Frame: up to 12 weeks after the last PDT, up to 24 weeks after first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions treated with narrow spectrum
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 39 | 125 | 126
Number analyzed (lesions treated with narrow spectrum) | 268 | 831 | 847
percentage of lesions | 32.5 [26.9 to 38.4] | 93.6 [91.7 to 95.2] | 89.3 [87.0 to 91.3]

22. Secondary Outcome: Change From Baseline in Total Lesion Area 3-4 Weeks After the First Photodynamic Therapy (PDT)
Description: Percentage of change from baseline in the lesion area of all treated lesions per subject (summation of sizes of all treated lesions) assessed at 3-4 weeks after the first PDT.
Time Frame: 3-4 weeks after the first PDT
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
percentage of change from baseline | -26.9 (32.74) | -78.9 (27.71) | -75.7 (27.76)

23. Secondary Outcome: Change From Baseline in Total Lesion Area 12 Weeks After the First Photodynamic Therapy (PDT)
Description: the change from baseline in the lesion area of all treated lesions per subject (summation of sizes of all treated lesions) assessed 12 weeks after the first PDT.
Time Frame: 12 weeks after the first PDT
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
percentage of change from baseline | -37.0 (39.86) | -85.4 (22.81) | -80.9 (27.65)

24. Secondary Outcome: Change From Baseline in Total Lesion Area 3-4 Weeks After the Second Photodynamic Therapy (PDT)
Description: the change from baseline in the lesion area of all treated lesions per subject (summation of sizes of all treated lesions) assessed 3-4 weeks after the second PDT. A second PDT was applied in case of non or partially responding lesions 12 weeks after first PDT.
Time Frame: 3-4 weeks after the second PDT, 15-16 weeks after first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 68 | 123 | 150
percentage of change from baseline | -46.2 (43.16) | -91.4 (15.83) | -87.5 (22.93)

25. Secondary Outcome: Change From Baseline in Total Lesion Area 12 Weeks After Second Photodynamic Therapy (PDT)
Description: the change from baseline in the lesion area of all treated lesions per subject (summation of sizes of all treated lesions) assessed 12 weeks after the second PDT. A second PDT was applied in case of non- or partially responding lesions 12 weeks after first PDT.
Time Frame: 12 weeks after the second PDT, 24 after first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 68 | 123 | 150
percentage of change from baseline | -50.1 (43.89) | -92.3 (17.15) | -88.9 (19.03)

26. Secondary Outcome: Change From Baseline in Total Lesion Area 3-4 Weeks After Last Photodynamic Therapy (PDT)
Description: the change from baseline in the lesion area of all treated lesions per subject (summation of sizes of all treated lesions) assessed at 3-4 weeks after last PDT, combining the changes from baseline in total lesion area of subjects 3-4 weeks after first PDT and second PDT (a second PDT was applied for subjects who showed non- or partially responding lesions 12 weeks after the first PDT).
Time Frame: 3-4 weeks after the last PDT, up to 16 weeks after the first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
percentage of change from baseline | -43.8 (43.40) | -89.4 (20.13) | -86.6 (22.57)

27. Secondary Outcome: Change From Baseline in Total Lesion Area 12 Weeks After Last Photodynamic Therapy (PDT)
Description: the change from baseline in the lesion area of all treated lesions per subject (summation of sizes of all treated lesions) assessed at 12 weeks after last PDT, combining the changes from baseline in total lesion area at 12 weeks after the first PDT and at 12 weeks after the second PDT (a second PDT was applied to subjects with non- or partially responding lesions 12 weeks after the first PDT).
Time Frame: 12 weeks after the last PDT, up to 24 weeks after the first treatment
Population: ITT
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
percentage of change from baseline | -48.5 (44.83) | -95.0 (15.66) | -92.0 (17.74)

28. Secondary Outcome: Overall Cosmetic Outcome of the Treated Skin 12 Weeks After Last Photodynamic Therapy (PDT) Compared to Baseline
Description: The cosmetic outcome 12 weeks after the last PDT (12 weeks after 1st PDT for subjects who are completely cleared at this time point, 12 weeks after 2nd PDT for subjects retreated due to remaining lesions 12 weeks after 1st PDT) will be calculated on the basis of the skin quality assessment (skin surface, hyperpigmentation, hypopigmentation, mottled or irregular pigmentation, degree of scarring, and atrophy) upon visual examination (scale: 0= none, 1= mild, 2= moderate, 3=severe). The cosmetic outcome is rated as very good if the sum score of the previously mentioned ratings (all ratings for each sign added up) has improved by at least 2 points as compared to baseline; as good if the sum score has improved by at least 1 point as compared to baseline; as satisfactory if the sum score is identical to the one at baseline; as unsatisfactory if the sum score has worsened by 1 point compared to baseline and as impaired if the sum score has worsened by at least 2 points compared to baseline.
Time Frame: 12 weeks after the last PDT, up to 24 weeks after first treatment
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 68 | 242 | 240
percentage of patients
  very good or good | 29.4 [19.0 to 41.7] | 36.0 [29.9 to 42.3] | 37.1 [31.0 to 43.5]
  very good | 14.7 [7.3 to 25.4] | 16.5 [12.1 to 21.8] | 19.2 [14.4 to 24.7]
  good | 14.7 [7.3 to 25.4] | 19.4 [14.6 to 25.0] | 17.9 [13.3 to 23.4]
  Satisfactory | 50.0 [37.6 to 62.4] | 55.8 [49.3 to 62.1] | 53.3 [46.8 to 59.8]
  Unsatisfactory | 16.2 [8.4 to 27.1] | 6.6 [3.8 to 10.5] | 5.8 [3.2 to 9.6]
  Impaired | 4.4 [0.9 to 12.4] | 1.7 [0.5 to 4.2] | 3.8 [1.7 to 7.0]

29. Secondary Outcome: Local Skin Reactions During First Photodynamic Therapy (PDT-1)
Description: Local skin reactions in the treatment area as assessed by the investigator during the first PDT (PDT-1)
Time Frame: during PDT treatment [3 h - 4 h ]
Population: Safety Population
Measure: Number; unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
percentage of patients
  Erythema | 32.9 | 72.6 | 71.1
  Edema | 1.3 | 22.2 | 23.6
  Induration | 0.0 | 9.3 | 8.5
  Vesicles | 0.0 | 3.2 | 6.1
  Erosion | 0.0 | 1.2 | 1.2
  Ulceration | 0.0 | 0.0 | 0.0
  Scaling/Flaking | 0.0 | 0.4 | 0.0
  Scabbing/Crusting | 0.0 | 0.4 | 0.0
  Weeping/Exudate | 0.0 | 0.4 | 1.2

30. Secondary Outcome: Local Skin Reactions During Second Photodynamic Therapy (PDT-2) for Retreated Subjects
Description: Local skin reactions in the treatment area as assessed by the investigator during PDT-2; only applicable for subjects who were retreated with a second PDT due to remaining lesions 12 weeks after the first PDT (subjects with data).
Time Frame: during PDT treatment [3 h - 4 h ]
Population: Safety Population - retreated subjects only
Measure: Number; unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 68 | 123 | 150
percentage of patients
  Erythema | 19.1 | 61.8 | 70.0
  Edema | 0.0 | 10.6 | 11.3
  Induration | 0.0 | 4.1 | 3.3
  Vesicles | 0.0 | 0.0 | 0.0
  Erosion | 0.0 | 0.0 | 0.0
  Ulceration | 0.0 | 0.0 | 0.0
  Scaling/Flaking | 0.0 | 0.0 | 0.0
  Scabbing/Crusting | 0.0 | 0.0 | 0.0
  Weeping/Exudate | 0.0 | 0.0 | 0.0

31. Secondary Outcome: Local Discomfort During First Photodynamic Therapy (PDT-1)
Description: Local discomfort reported by the patients during Illumination of first PDT (PDT1)
Time Frame: during PDT treatment [3 h - 4 h ]
Population: Safety Population
Measure: Number; unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
percentage of patients
  Itching during PDT-1 | 2.6 | 9.7 | 14.6
  Burning during PDT-1 | 28.9 | 81.9 | 85.8

32. Secondary Outcome: Local Discomfort During Second Photodynamic Therapy (PDT-2) for Retreated Subjects
Description: Local discomfort reported by the patients during Illumination phase of retreatment (PDT-2); only applicable for subjects who received a retreatment (PDT-2) due to remaining lesions 12 weeks after the first treatment (PDT-1) (subjects with data)
Time Frame: during PDT treatment [3 h - 4 h ]
Population: Safety Population - retreated subjects only
Measure: Number; unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 68 | 123 | 150
percentage of patients
  Itching during PDT-2 | 0.0 | 7.3 | 8.7
  Burning during PDT-2 | 14.7 | 69.9 | 74.7

33. Secondary Outcome: Local Discomfort - Pain During First Photodynamic Therapy (PDT-1)
Description: Pain (11-point numeric rating scale) by PDT Session; Overall (If both areas have been treated, maximum intensity over both areas is used for analysis.) Patients assessed the pain experienced during PDT using an 11-point numeric rating pain scale (NRPS) ranging from 0 (no pain at all) to 10 (worst possible pain). This score reflects the patient's maximum pain during PDT. This outcome measure shows pain score after the first PDT.
Time Frame: during PDT treatment [3 h - 4 h ]
Population: Safety Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
units on a scale | 0.5 (1.08) | 4.4 (3.50) | 4.4 (3.52)

34. Secondary Outcome: Local Discomfort - Pain During Second Photodynamic Therapy (PDT-2) for Retreated Subjects
Description: Pain (11-point numeric rating scale) by PDT Session; Overall (If both areas have been treated, maximum intensity over both areas is used for analysis.) Patients assessed the pain experienced during PDT using an 11-point numeric rating pain scale (NRPS) ranging from 0 (no pain at all) to 10 (worst possible pain). This score reflects the patient's maximum pain during PDT.
  Only applicable for subjects who received a retreatment (PDT-2) due to remaining lesions 12 weeks after the first treatment (PDT-1) (subjects with data)
Time Frame: during PDT treatment [3 h - 4 h ]
Population: Safety Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 68 | 123 | 150
units on a scale | 0.3 (1.10) | 3.1 (3.26) | 3.3 (3.22)

35. Secondary Outcome: Adverse Reactions
Description: Adverse reactions are Treatment-Emergent Adverse Events considered at least possibly related to the treatment with the randomized investigational medicinal products; Adverse reactions are shown with a frequency cut off of >=5%.
  TEAEs are considered from subjects who received only one PDT or subjects who received 2 PDTs (initial Treatment (PDT-1) and retreatment (PDT-2) due to remaining lesions 12 weeks after first photodynamic therapy.
  The safety set consists of all patients treated at least once with investigational product. Treatment with investigational product consists of application of study drug followed by illumination. This excludes one patient from the safety set; for this patient the investigational product was applied on the skin but it was not illuminated. Patients are treated according to actual treatment.
Time Frame: up to 12 weeks after the last PDT, up to 24 weeks after first treatment
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Number analyzed (Participants) | 76 | 248 | 246
Participants
  Application site irritation | 25 | 219 | 222
  Application site erythema | 31 | 198 | 199
  Application site pain | 19 | 175 | 179
  Application site edema | 1 | 62 | 61
  Application site pruritus | 6 | 59 | 60
  Application site exfoliation | 5 | 44 | 44
  Application site scab | 2 | 27 | 30
  Application site induration | 0 | 24 | 21
  Application site vesicles | 1 | 22 | 23
  Application site paraesthesia | 2 | 17 | 18
  Skin exfoliation | 1 | 17 | 15

ADVERSE EVENTS:
Time Frame: Until 12 weeks after the last treatment
Arm/Group | Vehicle | BF-200 ALA | MAL Cream
Serious Adverse Events (participants affected / at risk) | 3/76 | 11/248 | 10/246
Other Adverse Events (participants affected / at risk) | 55/76 | 239/248 | 241/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (N=76) | BF-200 ALA (N=248) | MAL Cream (N=246)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-Hodgkin's lymphoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Arterial stenosis limb (Vascular disorders) | 0 | 1 | 0
Temporal arteritis (Vascular disorders) | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (N=76) | BF-200 ALA (N=248) | MAL Cream (N=246)
Application site irritation (General disorders) | 25 | 219 | 222
Application site erythema (General disorders) | 31 | 198 | 199
Application site edema (General disorders) | 1 | 62 | 61
Application site pain (General disorders) | 19 | 175 | 179
Application site pruritus (General disorders) | 6 | 60 | 60
Application site exfoliation (General disorders) | 5 | 44 | 44
Application site scab (General disorders) | 2 | 27 | 30
Application site induration (General disorders) | 0 | 24 | 21
Application site vesicles (General disorders) | 1 | 22 | 23
Application site paraesthesia (General disorders) | 2 | 17 | 18
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 17 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The publication of study results requires Biofrontera's acceptance. Investigators can claim an authorship if they have completely treated and documented at least 35 patients. Planned publications and presentations of investigations which are within the scope of the clinical study should be previously presented to Biofrontera for a statement.